CLINICAL TRIAL: NCT07270692
Title: Detection of Reduced Left Ventricular Ejection Fraction With Three-Lead ECG Using Artificial Intelligence
Status: Recruiting | Type: Observational
Sponsor: Eko Devices, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2025.5
Record Dates: First submitted 2025-11-17; First posted 2025-12-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Low Ejection Fraction
Keywords: low ejection fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Eko digital stethoscopes — Use of the Eko CORE 500 digital stethoscope and 3M Littmann CORE Digital Stethoscope to auscultate and record cardiac phonocardiogram and (when available) electrocardiogram waveforms, as well as heart sounds.

SUMMARY:
The main objectives of this study are to train and evaluate an algorithm that predicts whether an individual has an ejection fraction ≤ 40%, using heart sounds and a 3-lead ECG as inputs, as well as determine the impact of gender, age, and race on algorithm performance.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Able and willing to provide informed consent
* Complete a clinical echocardiogram within 7 days before or after study procedures

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Patients who are hospitalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will employ an all-comers strategy, indicating that virtually any patient who receives a standard-of-care echocardiogram may participate. The echocardiogram must be within 7 days of the CORE 500 measurements to ensure that the measured ejection fraction is contemporaneous with the heart sounds and 3-lead ECG. This will include both healthy patients and patients with low EF.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Primary Objective: Collection of Heart Sounds and 3-lead ECG Recordings to Train Algorithm | 15-16 months
  The primary objective of this study is to train and evaluate an algorithm that predicts whether an individual has an ejection fraction ≤ 40%, by using Eko CORE 500 digital stethoscopes to collect the heart sounds and 3-lead ECG recordings of 500 patients who are 18 years or older and have completed an echocardiogram within 7 days of the study procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- P. D. Hinduja Hospital and Medical Research Centre, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No